CLINICAL TRIAL: NCT03390322
Title: DiaGone™ First in Human (FIH) Study - Safety and Performance of the DiaGone™ Device for the Treatment of Type 2 Diabetes
Brief Title: Safety and Initial Performance of the DiaGone Device on Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Digma Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLD-008
Record Dates: First submitted 2017-12-26; First posted 2018-01-04 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Duodenal Glycemic Control™ (Experimental)
  Interventions: Device: DiaGone™

INTERVENTIONS:
Device: DiaGone™ — Duodenal Glycemic Control™ using the DiaGone™ system

SUMMARY:
This is a multi-center, prospective, open label study of the Duodenal Glycemic Control™ procedure on type 2 diabetes patients sub-optimally controlled, to examine the safety and initial performance of the DiaGone™ system.

DETAILED DESCRIPTION:
This study is a multi-center, prospective, open label trial of type 2 diabetes patients sub-optimally controlled on at least one oral anti-diabetic medication.

Subjects who meet all inclusion and exclusion criteria after screening are hospitalized and go through the Duodenal Glycemic Control™ treatment.

Duodenal Glycemic Control™ treatment is conducted by a gastroenterologist, in an endoscopic suite, with an off-the-shelf endoscope, using the DiaGone™ system.

Patients are followed for 6 months for AE and SAE. Patients are followed for 12 months for glycemic control parameters.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are ≥ 18 years and ≤ 75 years of age.
* HbA1c at 7.5%-12%
* On oral glucose lowering drugs in a stable medication regimen
* Fasting plasma glucose level at ≥125mg/dL
* BMI 25-40 Kg/m2

Exclusion Criteria:

* Diagnosed Type I diabetes
* Serum C peptide <1ng/ml

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of procedure related SAEs. | 7 days
Incidence of procedure related SAEs. | 6 months

SECONDARY OUTCOMES:
Change to Fasting Glucose levels | 12 months
Change to Post Prandial Glucose levels | 12 months
Change to HbA1c levels | 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- IKEM, Prague, Czechia
- Israel (2):
  - Soroka Medical Center, Beersheba
  - Shaarei Tzedek, Jerusalem

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salinari S, Bertuzzi A, Guidone C, Previti E, Rubino F, Mingrone G. Insulin sensitivity and secretion changes after gastric bypass in normotolerant and diabetic obese subjects. Ann Surg. 2013 Mar;257(3):462-8. doi: 10.1097/SLA.0b013e318269cf5c. PMID 23388352
- [Background] Ferrannini E, Mingrone G. Impact of different bariatric surgical procedures on insulin action and beta-cell function in type 2 diabetes. Diabetes Care. 2009 Mar;32(3):514-20. doi: 10.2337/dc08-1762. No abstract available. PMID 19246589
- [Background] Mingrone G, Castagneto-Gissey L. Mechanisms of early improvement/resolution of type 2 diabetes after bariatric surgery. Diabetes Metab. 2009 Dec;35(6 Pt 2):518-23. doi: 10.1016/S1262-3636(09)73459-7. PMID 20152737
- [Background] de Jonge C, Rensen SS, Verdam FJ, Vincent RP, Bloom SR, Buurman WA, le Roux CW, Schaper NC, Bouvy ND, Greve JW. Endoscopic duodenal-jejunal bypass liner rapidly improves type 2 diabetes. Obes Surg. 2013 Sep;23(9):1354-60. doi: 10.1007/s11695-013-0921-3. PMID 23526068
- See also: Related Info — https://www.digmamedical.com